CLINICAL TRIAL: NCT05897073
Title: Impact of Time-Restricted Eating and Supervised Exercise on Hepatic Steatosis and Cardiometabolic Health in Adults With Obesity
Brief Title: Time-Restricted Eating, Exercise and Cardiometabolic Health in Obesity
Acronym: TEMPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEMPUS
Record Dates: First submitted 2023-05-05; First posted 2023-06-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Time Restricted Feeding; Exercise; Hepatic Steatosis; Cardiometabolic Syndrome; Obesity
MeSH Terms: conditions — Intermittent Fasting; Motor Activity; Fatty Liver; Metabolic Syndrome; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Time-restricted eating intervention (Experimental): Participants will be asked to reduce their daily eating time window to a maximum of 8 hours/day. They can choose when to begin their eating window but will be advised that the last meal should be completed before or at 20:00 hours. No calorie-containing food or beverage intake will be allowed outside the 8 hours eating window.
  Interventions: Behavioral: Time-restricted eating intervention
- Supervised exercise intervention (Experimental): The exercise intervention will include 2 days/week of supervised moderate-high intensity resistance training (rating perceived exertion >7, circuit-training, upper and lower body exercises involving major muscle groups) and high-intensity interval training (4 sets of 4-minute intervals at >85% peak heat rate with 4-minute of active recovery at 50-65% peak heat rate, uphill treadmill walking). Moreover, participants will receive an individualized moderate-intensity goal-setting aerobic (walking) program consisting of increasing 15% daily steps per week.
  Interventions: Behavioral: Exercise intervention
- Usual-care control group (No Intervention): Participants will receive standard recommendations on healthy lifestyle based on Mediterranean dietary pattern and physical activity recommendations for weight loss and health promotion.
- Time-restricted eating plus Supervised exercise (Experimental): Participants will be asked to reduce their daily eating time window to a maximum of 8 hours/day. They can choose when to begin their eating window but will be advised that the last meal should be completed before or at 20:00 hours. No calorie-containing food or beverage intake will be allowed outside the 8 hours eating window. The exercise intervention will include 2 days/week of supervised moderate-high intensity resistance training (rating perceived exertion >7, circuit-training, upper and lower body exercises involving major muscle groups) and high-intensity interval training (4 sets of 4-minute intervals at >85% peak heat rate with 4-minute of active recovery at 50-65% peak heat rate, uphill treadmill walking). Moreover, participants will receive an individualized moderate-intensity goal-
  Interventions: Behavioral: Time-restricted eating plus exercise intervention

INTERVENTIONS:
Behavioral: Time-restricted eating intervention — Participants will be asked to reduce their daily eating time window to a maximum of 8 hours/day. They can choose when to begin their eating window but will be advised that the last meal should be completed before or at 20:00 hours. No calorie-containing food or beverage intake will be allowed outside the 8 hours eating window.
  Arms: Time-restricted eating intervention
Behavioral: Exercise intervention — The exercise intervention will include 2 days/week of supervised moderate-high intensity resistance training (rating perceived exertion >7, circuit-training, upper and lower body exercises involving major muscle groups) and high-intensity interval training (4 sets of 4-minute intervals at >85% peak heat rate with 4-minute of active recovery at 50-65% peak heat rate, uphill treadmill walking). This intervention has already been tested previously in our lab. Moreover, participants will receive an individualized moderate-intensity goal-setting aerobic (walking) program consisting of increasing 15% daily steps per week.
  Arms: Supervised exercise intervention
Behavioral: Time-restricted eating plus exercise intervention — Participants will be asked to reduce their daily eating time window to a maximum of 8 hours/day. They can choose when to begin their eating window but will be advised that the last meal should be completed before or at 20:00 hours. No calorie-containing food or beverage intake will be allowed outside the 8 hours eating window. The exercise intervention will include 2 days/week of supervised moderate-high intensity resistance training (rating perceived exertion >7, circuit-training, upper and lower body exercises involving major muscle groups) and high-intensity interval training (4 sets of 4-minute intervals at >85% peak heat rate with 4-minute of active recovery at 50-65% peak heat rate, uphill treadmill walking). This intervention has already been tested previously in our lab. Moreover, participants will receive an individualized moderate-intensity goal-setting aerobic (walking) program consisting of increasing 15% daily steps per week.
  Arms: Time-restricted eating plus Supervised exercise

SUMMARY:
In Spain, overweight and obesity prevalence is reaching 70% in men and 50% in women. Excess of triglycerides are usually stored in the subcutaneous adipose tissue (SAT), until a point where SAT is unable to expand further. Therefore, lipids are deposited in visceral and other peripheral organs and tissues that are not otherwise designed for adipose storage such as the liver, pancreas or the skeletal muscle, a process known as ectopic fat deposition. "Time-restricted eating" (TRE) is a recently emerged intermittent fasting approach which has the potential to maximize the beneficial metabolic effects extensively reported for energy intake restriction. Furthermore, exercise reduces hepatic steatosis and improves cardiometabolic health in humans. However, whether the effects of TRE combined with exercise on reducing hepatic steatosis are superior to TRE or exercise intervention alone remains unknown. The TEMPUS study will investigate the effects of a 12-week TRE combined with supervised exercise intervention, as compared with TRE or exercise alone, and usual-care control group, on hepatic fat (primary outcome) and cardiometabolic health (secondary outcomes) in adults with obesity; and to unveil the role of gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25-65 years.
* Body mass index ≥28.0 and <40.0 kg/m2.
* Weight stability (within 5% of screening weight) for >3 months prior to study entry.
* Habitual eating window ≥11 hours.

Exclusion Criteria:

* History of a major adverse cardiovascular event, clinically significant kidney, endocrine, or neurological disease, bariatric surgery, HIV/AIDS, known inflammatory and/or rheumatologic disease, cancer, or other medical condition in which fasting or exercise is contraindicated.
* Type 1 or Type 2 diabetes.
* Major psychiatric disorders, eating disorders, sleep disorders, or alcohol abuse.
* Regular use of medication or compounds that may affect study outcomes (e.g., antidiabetic, steroids, beta-blockers, antibiotics, prebiotics, probiotics and symbiotics).
* Participating in a weight loss, a weight-management program or a supervised exercise program (more than 30 minutes three times per week, or 45 minutes twice a week, moderate/vigorous intensity).
* Pregnancy and lactation or planned pregnancy (within the study period).
* Caregiver for a dependent requiring frequent nocturnal care/sleep interruptions. Shift workers with variable hours (e.g., nocturnal).
* Frequent travel over time zones during the study period.
* Fear of needles and claustrophobia to magnetic resonance imaging (MRI).
* Being unable to understand and to accept the instructions or the study objectives and protocol.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Change in hepatic fat content | Change from baseline to 12 weeks
  Hepatic fat content will be assessed by Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Change in liver stiffness | Change from baseline to 12 weeks
  The quantification of stiffness will be assessed using attenuation imaging, shear wave elastography and shear wave dispersion with a Canon Aplio i800.
Change in values of alkaline phosphatase | Change from baseline to 12 weeks
  Fasting blood samples will be used to asses alkaline phosphatase
Change in values of alanine transaminase | Change from baseline to 12 weeks
  Fasting blood samples will be used to asses alanine transaminase
Change in values of gamma-glutamyl transferase | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess gamma-glutamyl transferase
Change in visceral adipose tissue | Change from baseline to 12 weeks
  Visceral adipose tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in abdominal subcutaneous adipose tissue | Change from baseline to 12 weeks
  Abdominal subcutaneous adipose tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in visceral adipose tissue | Change from baseline to 12 months
  Visceral adipose tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in abdominal subcutaneous adipose tissue | Change from baseline to 12 months
  Abdominal subcutaneous adipose tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in pancreatic fat content | Change from baseline to 12 weeks
  Pancreatic fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in pancreatic fat content | Change from baseline to 12 months
  Pancreatic fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in values of fasting glucose | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess glucose
Change in HOMA-IR index. | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess glucose and insulin and HOMA index will be computed
Change in values of HbA1c | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess HbA1c
Change in values of fasting triglycerides | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess levels of triglycerides
Change in values of fasting high-density lipoprotein cholesterol | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess levels of high-density lipoprotein cholesterol
Change in values of fasting low-density lipoprotein cholesterol | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess levels of low-density lipoprotein cholesterol
Change in values of fasting total cholesterol | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess levels of total cholesterol
Change in values of C-reactive protein | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess levels of C-reactive protein
Change in values of interleukin 6 | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess levels of interleukin 6
Change in values of apolipoprotein A1 | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess levels of apolipoprotein A1
Change in values of apolipoprotein B | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess levels of apolipoprotein B
Change in levels of mean glucose (Continuous Glucose Monitoring) | Change from baseline to the last 2 weeks of intervention
  24-hour, diurnal and nocturnal mean glucose over 14 days will be assessed by Continuous Glucose Monitoring during 2 weeks
Change in 2-hour plasma glucose | Change in 2-hour plasma glucose baseline and 12 weeks
  2-hour plasma glucose will be assessed by oral glucose tolerance test.
Change in Body weight | Change from baseline to 12 weeks
  Body weight will be measured by a digital scale
Change in Body weight | Change from baseline to 12 months
  Body weight will be measured by a digital scale
Change in Body height | Change from baseline to 12 weeks
  Body height will be measured by a stadiometer
Change in Body height | Change from baseline to 12 months
  Body height will be measured by a stadiometer
Change in waist circumference | Change from baseline to 12 weeks
  Waist circumference will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in calf girth | Change from baseline to 12 weeks
  Calf girth will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in waist circumference | Change from baseline to 12 months
  Waist circumference will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in calf girth | Change from baseline to 12 months
  Calf girth will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in hip circumference | Change from baseline to 12 weeks
  Hip circumference will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in hip circumference | Change from baseline to 12 months
  Hip circumference will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in neck circumference | Change from baseline to 12 weeks
  Neck circumference will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in neck circumference | Change from baseline to 12 months
  Neck circumference will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in systolic blood pressure | Change from baseline to 12 weeks
  Systolic blood pressure will be assessed by blood pressure monitor
Change in systolic blood pressure | Change from baseline to 12 months
  Systolic blood pressure will be assessed by blood pressure monitor
Change in diastolic blood pressure | Change from baseline to 12 weeks
  Diastolic blood pressure will be assessed by blood pressure monitor
Change in diastolic blood pressure | Change from baseline to 12 months
  Diastolic blood pressure will be assessed by blood pressure monitor
Change in energy intake | Change from baseline to 12 weeks
  Energy intake (kcal/day) will be assessed by 24h recalls
Change in carbohydrates intake | Change from baseline to 12 weeks
  Macronutrients intake (g/day and percentage of energy intake) will be assessed by 24h recalls
Change in fat intake | Change from baseline to 12 weeks
  Fat intake (g/day and percentage of energy intake) will be assessed by 24h recalls
Change in protein intake | Change from baseline to 12 weeks
  Protein intake (g/day and percentage of energy intake) will be assessed by 24h recalls
Change in dietary habits | Change from baseline to 12 weeks
  Dietary habits will be assessed by food frequency questionnaire (FFQ). Minimum value is 1 (never) and maximum value is 9 (more than 6 times per day). Higher values mean a more frequency of a certain food consumption.
Change in Appetite traits | Change from baseline to 12 weeks
  Appetite traits will be assessed by the Adult Eating Behavior Questionnaire (AEBQ). Minimum value is 1 (completely disagree) and maximum value is 5 (completely agree). Higher values mean a worse outcome.
Change in Subjective sleep quality | Change from baseline to 12 weeks
  Subjective sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI). Minimum value is 0 (never) and maximum value is 3 (3 or more times per week). Higher values mean a worse outcome.
Change in Objectively sleep quality | Change from baseline to 12 weeks
  Objectively sleep quality will be assessed by accelerometry
Change in Chronotype | Change from baseline to 12 weeks
  Chronotype will be assessed by the Munich Chronotype Questionnaire (MCTQ).
Change in Morning-Evening type | Change from baseline to 12 weeks
  Morning-Evening type will be assessed by the Morningness-Eveningness Questionnaire Self-Assessment Version. Define if a person is more morningness or eveningness based on daily times preferences.
Change Objectively moderate to vigorous physical activity levels | Change from baseline to 12 weeks
  Objectively physical activity levels will be assessed by accelerometry
Change in Depression aspects | Change from baseline to 12 weeks
  Depression aspects will be assessed by the Beck Depression Inventory Fast Screen (BDI-FS). Values ranged from 0 to 63. Higher values mean worse outcome.
Change in Stress aspects | Change from baseline to 12 weeks
  Stress aspects will be assessed by the Perceived Stress Scale (PSS). Values ranged from 0 to 40. Higher values mean worse outcome.
Change in Anxiety aspects | Change from baseline to 12 weeks
  Anxiety aspects will be assessed by the State-Trait Anxiety Inventory (STAI). Values ranged from 0 to 60. Higher values mean worse outcome.
Change in General health | Change from baseline to 12 weeks
  General health will be assessed by the EuroQol 5 dimensions 5 levels (EQ-5D-5L). Values ranged from 0 to 100. Higher values mean better outcome.
Change in Quality of life | Change from baseline to 12 weeks
  Quality of life will be assessed by the Rand Short Form 36 (SF-36). Values ranged from 0 to 100. Higher values mean better outcome.
Change in fecal microbiota composition | Change from baseline to 12 weeks
  Shotgun metagenomic sequencing of DNA extracted from stool samples to determine taxonomic profiling (e.g., phylum, genera, species).
Change in fecal microbiota diversity | Change from baseline to 12 weeks
  Shotgun metagenomic sequencing of DNA extracted from stool samples to determine fecal microbiota diversity (e.g., beta and alpha diversity metrics).
Change in Cardiorespiratory Fitness | Change from baseline to 12 weeks
  Cardiorespiratory fitness measured by maximum treadmill test
Change in Lower muscular strength | Change from baseline to 12 weeks
  Lower body muscular strength measured by chair stand test.
Change in Upper muscular strength | Change from baseline to 12 weeks
  Upper body muscular strength measured by hand grip strength test.
Change in walking speed. | Change from baseline to 12 weeks
  Walking speed measured by gait speed test. Higher values mean worse performance.
Adherence to the eating window | During the 12 weeks
  Adherence will be assessed by eating records through the mobile phone app.
Attendance to the exercise intervention | During the 12 weeks
  Attendance will be assessed by number of completed exercise sessions.
Change in hepatic fat content | Change from baseline to 12 months
  Hepatic fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in abdominal intermuscular fat content | Change from baseline to 12 weeks
  Abdominal intermuscular fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in abdominal intermuscular fat content | Change from baseline to 12 months
  Abdominal intermuscular fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in abdominal skeletal muscle tissue | Change from baseline to 12 months
  Abdominal skeletal muscle tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in abdominal skeletal muscle tissue | Change from baseline to 12 weeks
  Abdominal skeletal muscle tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in mid-thigh subcutaneous adipose tissue | Change from baseline to 12 weeks
  Mid-thigh subcutaneous adipose tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in mid-thigh subcutaneous adipose tissue | Change from baseline to 12 months
  Mid-thigh subcutaneous adipose tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in mid-thigh intermuscular fat content | Change from baseline to 12 weeks
  Mid-thigh intermuscular fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in mid-thigh intermuscular fat content | Change from baseline to 12 months
  Mid-thigh intermuscular fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in mid-thigh intramuscular fat content | Change from baseline to 12 weeks
  Mid-thigh intramuscular fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in mid-thigh intramuscular fat content | Change from baseline to 12 months
  Mid-thigh intramuscular fat content will be assessed by Magnetic Resonance Imaging (MRI)
Change in mid-thigh skeletal muscle tissue | Change from baseline to 12 weeks
  Mid-thigh skeletal muscle tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in mid-thigh skeletal muscle tissue | Change from baseline to 12 months
  Mid-thigh skeletal muscle tissue will be assessed by Magnetic Resonance Imaging (MRI)
Change in liver stiffness | Change from baseline to 12 months
  The quantification of stiffness will be assessed using attenuation imaging, shear wave elastography and shear wave dispersion with a Canon Aplio i800.
Change in liver steatosis | Change from baseline to 12 weeks
  The quantification of steatosis will be assessed using attenuation imaging, shear wave elastography and shear wave dispersion with a Canon Aplio i800.
Change in liver steatosis | Change from baseline to 12 months
  The quantification of steatosis will be assessed using attenuation imaging, shear wave elastography and shear wave dispersion with a Canon Aplio i800.
Change in liver viscosity | Change from baseline to 12 weeks
  The quantification of viscosity will be assessed using attenuation imaging, shear wave elastography and shear wave dispersion with a Canon Aplio i800.
Change in liver viscosity | Change from baseline to 12 months
  The quantification of viscosity will be assessed using attenuation imaging, shear wave elastography and shear wave dispersion with a Canon Aplio i800.
Change in Fat Mass | Change from baseline to 12 weeks
  Fat mass will be assessed by assessed by bioelectrical impedance analysis (BIA).
Change in Fat Mass | Change from baseline to 12 months
  Fat mass will be assessed by assessed by bioelectrical impedance analysis (BIA).
Change in Fat-free Mass | Change from baseline to 12 weeks
  Fat-free mass will be assessed by assessed by bioelectrical impedance analysis (BIA).
Change in Fat-free Mass | Change from baseline to 12 months
  Fat-free mass will be assessed by assessed by bioelectrical impedance analysis (BIA).
Change in Bone Mineral Density | Change from baseline to 12 months
  Bone mineral density will be assessed by dual-energy X-ray absorptiometry scans (DXA).
Change in Bone Mineral Density | Change from baseline to 12 weeks
  Bone mineral density will be assessed by dual-energy X-ray absorptiometry scans (DXA).
Change in values of alkaline phosphatase | Change from baseline to 12 months
  Fasting blood samples will be used to asses alkaline phosphatase
Change in values of alanine transaminase | Change from baseline to 12 months
  Fasting blood samples will be used to asses alanine transaminase
Change in values of aspartate aminotransferase | Change from baseline to 12 weeks
  Fasting blood samples will be used to asses aspartate aminotransferase
Change in values of aspartate aminotransferase | Change from baseline to 12 months
  Fasting blood samples will be used to asses aspartate aminotransferase
Change in values of gamma-glutamyl transferase | Change from baseline to 12 months
  Fasting blood samples will be used to assess gamma-glutamyl transferase
Change in values of HbA1c | Change from baseline to 12 months
  Fasting blood samples will be used to assess HbA1c
Change in values of fasting glucose | Change from baseline to 12 months
  Fasting blood samples will be used to assess glucose
Change in values of fasting insulin | Change from baseline to 12 weeks
  Fasting blood samples will be used to assess insulin
Change in values of fasting insulin | Change from baseline to 12 months
  Fasting blood samples will be used to assess insulin
Change in HOMA-IR index. | Change from baseline to 12 months
  Fasting blood samples will be used to assess glucose and insulin and HOMA index will be computed
Change in values of fasting triglycerides | Change from baseline to 12 months
  Fasting blood samples will be used to assess levels of triglycerides
Change in values of fasting high-density lipoprotein cholesterol | Change from baseline to 12 months
  Fasting blood samples will be used to assess levels of high-density lipoprotein cholesterol
Change in values of fasting low-density lipoprotein cholesterol | Change from baseline to 12 months
  Fasting blood samples will be used to assess levels of low-density lipoprotein cholesterol
Change in values of fasting total cholesterol | Change from baseline to 12 months
  Fasting blood samples will be used to assess levels of total cholesterol
Change in values of apolipoprotein A1 | Change from baseline to 12 months
  Fasting blood samples will be used to assess levels of apolipoprotein A1
Change in values of apolipoprotein B | Change from baseline to 12 months
  Fasting blood samples will be used to assess levels of apolipoprotein B
Change in values of C-reactive protein | Change from baseline to 12 months
  Fasting blood samples will be used to assess levels of C-reactive protein
Change in values of interleukin 6 | Change from baseline to 12 months
  Fasting blood samples will be used to assess levels of interleukin 6
Change in values of essential amino acids | Change from baseline to 12 weeks
  Fasting urine samples will be used to assess levels of essential amino acids.
Change in values of non-essential amino acids | Change from baseline to 12 weeks
  Fasting urine samples will be used to assess levels of essential amino acids.
Change in fiber intake | Change from baseline to 12 weeks
  Fiber intake (g/day and percentage of energy intake) will be assessed by 24h recalls
Change in rest-activity rhythms | Change from baseline to the last 2 weeks of intervention
  Rest-activity rhythms will be assessed by accelerometry
Change in steps counts | Change from baseline to the last 2 weeks of intervention
  Steps counts will be assessed by activity band
Change in Fat Mass | Change from baseline to 6 weeks
  Fat mass will be assessed by assessed by bioelectrical impedance analysis (BIA).
Change in Fat-free Mass | Change from baseline to 6 weeks
  Fat-free mass will be assessed by assessed by bioelectrical impedance analysis (BIA).
Change in Body weight | Change from baseline to 6 weeks
  Body weight will be measured by a digital scale
Change in waist circumference | Change from baseline to 6 weeks
  Waist circumference will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in hip circumference | Change from baseline to 6 weeks
  Hip circumference will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in neck circumference | Change from baseline to 6 weeks
  Neck circumference will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in calf girth | Change from baseline to 6 weeks
  Calf girth will be assessed by measuring tape following the procedures outlined by the International Society for the Advancement of Kinanthropometry
Change in Bone Mineral Density | Change from baseline to 6 weeks
  Bone mineral density will be assessed by dual-energy X-ray absorptiometry scans (DXA).
Change in fecal microbiota functionality | Change from baseline to 12 weeks
  Shotgun metagenomic sequencing of DNA extracted from stool samples to determine microbial functional capacity through the analysis of metabolic pathways.
Change in fiber intake | Change from baseline to 6 weeks
  Fiber intake (g/day and percentage of energy intake) will be assessed by 24h recalls
Change in carbohydrates intake | Change from baseline to 6 weeks
  Macronutrients intake (g/day and percentage of energy intake) will be assessed by 24h recalls
Change in protein intake | Change from baseline to 6 weeks
  Protein intake (g/day and percentage of energy intake) will be assessed by 24h recalls
Change in energy intake | Change from baseline to 6 weeks
  Energy intake (kcal/day) will be assessed by 24h recalls
Change in fat intake | Change from baseline to 6 weeks
  Fat intake (g/day and percentage of energy intake) will be assessed by 24h recalls
Change in adherence to Mediterranean diet | Change from baseline to 6 weeks
  Adherence to the Mediterranean dietary pattern will be assessed using validated questionnaires such as the PREDIMED questionnaire. The minimum value is 0 and the maximum value is 14. Higher values indicate better adherence to the Mediterranean diet and represent a better outcome.
Change in adherence to Mediterranean diet | Change from baseline to 12 weeks
  Adherence to the Mediterranean dietary pattern will be assessed using validated questionnaires such as the PREDIMED questionnaire. The minimum value is 0 and the maximum value is 14. Higher values indicate better adherence to the Mediterranean diet and represent a better outcome.
Change in adherence to Mediterranean diet | Change from baseline to 12 months
  Adherence to the Mediterranean dietary pattern will be assessed using validated questionnaires such as the PREDIMED questionnaire. The minimum value is 0 and the maximum value is 14. Higher values indicate better adherence to the Mediterranean diet and represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan R. Ruiz, PhD, Principal Investigator — Universidad de Granada
Locations (2):
- Spain (2):
  - University of Granada - Instituto Mixto Universitario Deporte y Salud, Granada, Granada
  - University of Granada, Granada, Granada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camacho-Cardenosa A, Clavero-Jimeno A, Martin-Olmedo JJ, Amaro-Gahete F, Cupeiro R, Cejudo MTG, Garcia Perez PV, Hernandez-Martinez C, Sevilla-Lorente R, De-la-O A, Lopez-Vazquez A, Molina-Fernandez M, Carneiro-Barrera A, Garcia F, Rodriguez-Nogales A, Galvez Peralta JJ, Cabeza R, Martin-Rodriguez JL, Munoz-Garach A, Munoz-Torres M, Labayen I, Ruiz JR. Time-restricted eating and supervised exercise for improving hepatic steatosis and cardiometabolic health in adults with obesity: protocol for the TEMPUS randomised controlled trial. BMJ Open. 2024 Jan 24;14(1):e078472. doi: 10.1136/bmjopen-2023-078472. PMID 38267239

DOCUMENTS (2):
  • Study Protocol (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05897073/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05897073/SAP_001.pdf